CLINICAL TRIAL: NCT07022197
Title: Safety and Efficacy of BAFF-R CART for Refractory Neuroimmune Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Liu, Department of Neurology, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB2024-YX-274-01
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy; NMO Spectrum Disorder; Myasthenia Gravis; Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Neuromyelitis Optica; Myasthenia Gravis; Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group BAFF-R CART cells (Experimental): Experimental: CART cells therapy，Dose level 1: 0.5 × 10^6 CART cells/Kg The tolerability and safety of BAFF-R CART cells will be assessed in an initial dose of 0.5×10^6 CART cells/Kg and three subjects will be enrolled firstly.
  Experimental: CART cells therapy，Dose level 2: 1 × 10^6 CART cells/Kg If neither DLT nor efficacy is shown in the first three subjects, the dose of CART cells will be increased to 1 × 10^6 CART cells/kg to assess DLT.
  Experimental: CART cells therapy，Dose level 3: 2 × 10^6 CART cells/Kg If DLT occurs in two subjects, whether to test the safety and efficacy in 2 × 10^6 CART cells/kg group will be determined by the investigator based on the initial data of efficacy, PK and PD.
  Interventions: Drug: BAFF-R CART

INTERVENTIONS:
Drug: BAFF-R CART — Biological: BAFF-R CART cells Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to manufacture BAFF-R CART cells, during which cyclophosphamide will be administered for the purpose of lymphocytes depletion. After lymphodepletion, subjects will receive one dose treatment with BAFF-R CART cells by intravenous (IV) infusion. The initial dose of 0.5×10^6 CART cells/kg will be infused on day 0.
  Drug: Cyclophosphamide and fludarabine Subjects will receive one 3-day cycle of lymphodepletion starting 4 days prior to BAFF-R CART cells infusion on Day 0.
  Subjects will be given IV infusion of cyclophosphamide 250 mg/m2/day on day -5, -4 and -3, and fludarabine 30 mg/m2 over 30 minutes administered immediately after cyclophosphamide.

SUMMARY:
This study is a phase Ib/IIa dose-escalation study designed to evaluate the safety, tolerability, and preliminary efficacy of autologous T cells expressing chimeric antigen receptor (CAR)-targeted B-cell activating factor receptor (BAFFR) in refractory neuroimmune diseases. The study design is divided into two parts, the first of which will be given to each patient at 3 incremental dose levels to establish the maximum tolerated dose (MTD). Each disease is expected to enroll 12 patients who meet the inclusion criteria. In the second part, 15 patients per disease will be recruited to further characterize the efficacy of the MTD.

DETAILED DESCRIPTION:
* Phase I: Frequency, type, and severity of adverse events (according to the National Cancer Institute Common Terminology Criteria for Adverse Events CTCAE V5.0) occurring within 4 weeks after BAFF-R CART infusion;
* Phase II: Number of recurrences at 52 weeks after BAFF-R CART infusion;
* Characterization of BAFF-R CART cell expansion levels over time in subjects (peripheral blood, cerebrospinal fluid, bone marrow, etc.);
* Characteristics of BAFF-R+ B cell and antibody secreting cell (ASC) lymphocyte ablation in subjects;
* Changes in disease-related clinical scores at baseline, 24 and 52 weeks after BAFF-R CART infusion;
* Changes in the cumulative total number of MRI active lesions in MS and NMOSD patients at 24 and 52 weeks after BAFF-R CART infusion;
* Frequency, type, and severity of treatment-related laboratory index abnormalities (according to the National Cancer Institute Common Terminology Criteria for Adverse Events CTCAE V5.0);
* Characterization of changes in disease-associated antibody titers in the subject;
* Changes in vital signs (blood pressure, pulse rate, weight, ECG).

ELIGIBILITY:
Inclusion Criteria:

1. Assessed by the investigator as having a refractory neuroimmune disease;

Refractory neuroimmune diseases were defined as:

1. Poor symptom control on at least three immunosuppressive agents for more than one year;
2. Clinical evidence of at least two relapses within 12 months or three relapses within 24 months and one relapse within 12 months prior to screening.

2. Male study participants must agree to use contraception during the treatment period for 1 year after receiving study treatment, and sperm donation is prohibited throughout the study period;

3. In the case of females with childbearing potential, need to agree to use contraception during the treatment period and for at least 1 year after receiving study treatment. Participants must have a negative serum pregnancy test result at screening and a confirmed negative urine pregnancy test result prior to first CART treatment.

Exclusion Criteria:

1. Any medical or psychiatric condition that, in the opinion of the investigator, may jeopardize the study participant or affect the study participant's ability to participate in this study;
2. A history of drug or alcohol abuse within the 12 months prior to baseline, or any condition that in the opinion of the investigator is associated with poor adherence;
3. Women who are breastfeeding or pregnant, or who plan to become pregnant at any time during the 12-month time period following treatment with CART, or a history of spontaneous or induced abortion within 4 weeks prior to screening;
4. Study participants with a clinically relevant active infection (e.g., sepsis, pneumonia, or abscess) or serious infection (resulting in hospitalization or requiring antibiotic therapy) within 4 weeks prior to baseline;
5. The study participant has received a live attenuated vaccination within 8 weeks prior to baseline; or is scheduled to receive a live vaccination (including COVID-19 vaccine) within 8 weeks after treatment;
6. Study participants who have received prior treatment with rituximab within 6 months prior to baseline;
7. Study participants had received tolizumab, eculizumab within 3 months prior to baseline;
8. Study participants who have received intravenous human immunoglobulin, plasma exchange, undergone immunotherapy within 4 weeks prior to baseline;
9. Known concomitant serious underlying diseases, such as hepatic and renal impairment, hematologic disorders, previous severe cardiovascular disease, severe hypertension, diabetes mellitus, poor control of blood pressure and blood glucose;
10. Comorbid mental illness, suicidal ideation (affirmative answer (yes) to question 4 or question 5 of the Colombian Suicide Severity Rating Scale (C-SSRS) indicating a suicide attempt within the last 6 months);
11. Any of the following laboratory abnormalities during the screening period (a repeat measurement may be taken during the screening period prior to randomization to confirm results); (1) Elevated liver enzymes: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal (ULN); (2) Total bilirubin > 1.5 times the ULN; (3) Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2; (4) CD19 + B cell count <40 cells/µL;
12. Presence of a history of tuberculosis infection, high risk of acquired tuberculosis infection;
13. known immunodeficiency diseases, including human immunodeficiency virus (HIV) infection;
14. Viral hepatitis B surface antigen (HBsAg) positivity during the screening period;
15. Receiving blood transfusion therapy 4 weeks prior to baseline or during the screening period;
16. Any other condition that the investigator deems inappropriate for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Types and incidence of dose-limiting toxicity (DLT) after BAFF-R CART cells infusion | Up to 3 months post BAFF-R CART cells infusion
  To evaluate the DLT occurred within 3 months after BAFF-R CART cells infusion.
Incidence and severity of AEs, including changes in vital signs, physical examination, laboratory parameters, Electrocardiograms and Echocardiograms. | Up to 2 years post BAFF-R CART cells infusion
  To evaluate the AEs occurred within 2 years after BAFF-R CART cells infusion.

SECONDARY OUTCOMES:
PD-Soluble BAFF | Up to 2 years post BAFF-R CART cells infusion
  The changes of concentration of soluble BAFF in the peripheral blood after BAFF-R CART cells infusion.
PD-Pathogenic antibody | Up to 2 years post BAFF-R CART cells infusion
  The changes of pathogenic antibody titers in peripheral blood or cerebrospinal fluid.
PD-Nfl（MS） | Up to 2 years post BAFF-R CART cells infusion
  The changes of peripheral blood Neurofilament Light chain (NfL) concentration in patients with MS.
PK-VCN | Up to 15 years post BAFF-R CART cells infusion
  The number of BAFF-R CAR gene copies (VCN, copies/μg DNA) in peripheral blood and cerebrospinal fluid after administration.
PK-BAFF-R CAR-T cells | Up to 2 years post BAFF-R CART cells infusion
  The concentration of BAFF-R CAR T cells (cells/mL) in peripheral blood after administration was detected by flow cytometry.

OTHER OUTCOMES:
NMOSD: the number of attacks | Up to 2 years post BAFF-R CART cells infusion
  The number of attacks divided by observed year after BAFF-R CART cells infusion.
NMOSD: Accumulated total active MRI lesions | Up to 2 years post BAFF-R CART cells infusion
  the number of accumulate total active MRI lesions after BAFF-R CART cells infusion.
NMOSD: Expanded Disability Status Scale (EDSS) score | Up to 2 years post BAFF-R CART cells infusion
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS). It consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline indicates improvement. A participant was considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.
NMOSD: Modified Rankin Scale | Up to 2 years post BAFF-R CART cells infusion
  Modified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. We characterized a favorable outcome as mRS ranging from zero up to two, while unfavorable outcome ranging for 3 up to 6.
NMOSD: Visual acuity | Up to 2 years post BAFF-R CART cells infusion
  Corrected visual acuity is determine by Snellen E chart held at a distance of 5 meters. Higher score indicates better vision.
MG: Quantitative Myasthenia Gravis Score (QMG) | Up to 2 years post BAFF-R CART cells infusion
  The QMG score is a 13-item scale used to quantify disease severity in myasthenia gravis. The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).
MG: Myasthenia Gravis Activities if Daily Living (MG-ADL) Score | Up to 2 years post BAFF-R CART cells infusion
  The MG-ADL is an eight-question survey of symptom severity, with each response graded from 0 (normal) to 3 (most severe). Two questions concern ocular, three oropharyngeal, one respiratory, and two extremity functions. Cumulative MG-ADL scores range from 0 to 24.
CIDP: Inflammatory Neuropathy Cause and Treatment (INCAT) Score | Up to 2 years post BAFF-R CART cells infusion
  The INCAT score comprises two parts, the arm score and the leg score. Based on a patient's level of impairment in their arms and legs, each part is scored between 0 and 5 points, resulting in an INCAT total score between 0 and 10.
CIDP: Medical Research Council (MRC) muscle function Score | Up to 2 years post BAFF-R CART cells infusion
  The MRC score system for testing and grading of muscle function aims to provide a standardized and objective way to assess muscle function. It ranges from 0 to 5.
CIDP: Assess changes in nerve conduction test results | Up to 2 years post BAFF-R CART cells infusion
  Including motor nerve distal latency, proximal latency, compound muscle motor potential (CMAP), motor nerve conduction velocity, sensory nerve conduction velocity, sural nerve potential.
IMNM: Manual Muscle Testing (MMT) Score | Up to 2 years post BAFF-R CART cells infusion
  For MMT score, 16 muscle groups/ motions will be tested (not individual muscles). 14 of these are tested bilaterally.
IMNM: Assess the changes in serum creatine kinase levels in patients with IMNM before and after treatment. | Up to 2 years post BAFF-R CART cells infusion
  If the creatine kinase level drops to twice the upper limit of normal or below, it is defined as effective, and the effective rate is calculated.
IMNM: Muscle MRI | Up to 2 years post BAFF-R CART cells infusion
  Calculating the hyperintensity of muscle MRI T2/STIR sequence in patients with IMNM.
36-item Short Form Generic Health Survey (SF-36) score | Up to 2 years post BAFF-R CART cells infusion
  SF-36 will used to understand the health related quality-of -life of the subjects after BAFF-R CART cells infusion. The eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions will be searched. These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.
EuroQol-five dimensions (EQ-SD) score | Up to 2 years post BAFF-R CART cells infusion
  Health status is measured with the EuroQuality of Life Five Dimensions (EQ-5D) after BAFF-R CART cells infusion, which includes five dimensions and is used to evaluate the quality of life of sepsis survivors. They are mobility, self-care, usual activities, discomfort or pain and depression or anxiety. Levels are coded 1-5 and a total score is then generated. Results for the demographic measured will be displayed as a percentage value.
Visual analogue scale (VAS) pain score | Up to 2 years post BAFF-R CART cells infusion
  usual visual analog scale (VAS) of pain is used to evaluate pain after BAFF-R CART cells infusion (line from 0: no pain to 10:worst pain).
Annual hospitalization rates | Up to 2 years post BAFF-R CART cells infusion
  The number of In-patient hospitalization is defined as a stay in hospital that goes beyond midnight of the first day of admission.
Cytokines release after BAFF-R CART cells infusion | Up to 2 years post BAFF-R CART cells infusion
  Changes of concentration( pg/mL) of cytokines ( such as ferritin, CRP, IL-6 and procalcitonin) will be analyzed after Changes of concentration( pg/mL) of cytokines ( such as ferritin, CRP, IL-6 and procalcitonin) will be analyzed after BAFF-R CART cells infusion.
Immunogenicity of BAFF-R CART cells | Up to 2 years post BAFF-R CART cells infusion
  Anti-drug antibodies (ADA) against CAR on BAFF-R CART cells will be analyzed after BAFF-R CART cells infusion.
Detection of RCL | Up to 2 years post BAFF-R CART cells infusion
  Levels of replication competent lentivirus (RCL) will be monitored after BAFF-R CART cells infusion.
Profiling of cell subtypes | Up to 2 years post BAFF-R CART cells infusion
  Changes in cells in infused CART products, blood and CSF (including proportion of CD3+ T cells, CD3+CD4+ T cells and CD3+CD8+ T cells, ratio of CD4+ T/CD8+T, and single-cell sequencing) will be analyzed after BAFF-R CART cells infusion.
MS: Annualized Relapse Rate (ARR) | Up to 2 years post BAFF-R CART cells infusion
  Annualized relapse rate (ARR): Number of MS relapses divided by observed year after BAFF-R CART cells infusion.
MS: Time to first relapse | Up to 2 years post BAFF-R CART cells infusion
  Time from BAFF-R CART cells infusion to the first relapse of MS.
MS: Number of T1 Gadolinium (Gd) | Up to 2 years post BAFF-R CART cells infusion
  The changes of enhancing Lesions as detected by brain Magnetic Resonance Imaging (MRI).
MS: Annualized rate of T2 lesions | Up to 2 years post BAFF-R CART cells infusion
  Annualized rate of T2 lesions：Number of New, and/or Enlarging T2 Hyperintense Lesions as detected by MRI divided by observed year after BAFF-R CART cells infusion.
MS: Percent Change in T2 lesions volume | Up to 2 years post BAFF-R CART cells infusion
  The percent change of T2 lesions volume as detected by MRI from the baseline.
MS: Change in EDSS | Up to 2 years post BAFF-R CART cells infusion
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS).
MS: Percent of NEDA-3 | Up to 2 years post BAFF-R CART cells infusion
  The no evidence of disease activity-3 (NEDA-3), defined as no relapse, no disability worsening, and no MRI activity.
MS: 3-month CDP | Up to 3 months post BAFF-R CART cells infusion
  Time to onset of 3-month CDP as assessed by EDSS score.
MS: 6-month CDP | Up to 6 months post BAFF-R CART cells infusion
  Time to onset of 6-month CDP as assessed by EDSS score.
MS: Patient Reported Outcomes (PRO) | Up to 2 years post BAFF-R CART cells infusion
  Including Fatigue Symptoms and Impacts Questionnaire -Relapsing Multiple Sclerosis (FSIQ-RMS), General Anxiety Disorder Scale (GAD-7), Patient Health Questionnaire (PHQ-9), Health Utilities Index (HUI-III), Multiple Sclerosis Impact Scale (MSIS-29).

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, M.D.,Ph.D, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China